CLINICAL TRIAL: NCT00066040
Title: Prevention of Transmission of Mutans Streptococci From Mother to Child
Brief Title: Prevention of Transmission of Bacteria That Cause Cavities From Mothers to Their Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDCR-13534; R01DE013534 (NIH); NCT00016822 (obsolete NCT alias)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2012-07

CONDITIONS: Caries, Dental
Keywords: mutans streptococci infections
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cervitec chlorhexidine varnish
Drug: Duraphat fluoride varnish
Drug: xylitol gum from Fennobon, Finland

SUMMARY:
The purpose of this study is to control the levels of bacteria that causes cavities in mothers by a combination of treatments that include fluoride and chlorhexidine varnishes and xylitol-chewing gum before the appearance of teeth in the mouth of their children. By doing that we expect to reduce the acquisition of the bacteria that causes cavities (the mutans streptococci) by the children which in turn will reduce the development of cavities.

DETAILED DESCRIPTION:
Dental decay is the most prevalent affliction in children worldwide. In recent years the occurrence of dental decay has declined dramatically in many industrialized countries subsequent to the widespread availability of fluoride in the water supply and dentifrices. However, in newly industrialized countries such as Brazil, the occurrence of decay is still high, especially among lower income groups. The mutans streptococci (MS) have been convincingly associated with human dental decay and clinical protocols, which seek to reduce the levels of MS invariably, thus resulting in a significant reduction in decay. One of the most important observations from these studies is the possibility that decay and the establishment of MS can be reduced and/or prevented in young children by treating those mothers who are highly infected with MS prior to the eruption of the primary teeth. Other studies indicate that if the MS does not colonize the primary teeth in the first year after their eruption, they are likely to remain caries free during the following years. These findings indicate that delaying the colonization of the MS in the primary dentition may prevent dental decay. The ideal population for such a study can be found in communities without water fluoridation, with a high level of unmet dental care, and who would have frequent access to sugar. Populations in many newly industrialized countries would meet these qualifications. However, it is difficult to perform an interceptive study, such as preventing the transmission of the MS from mother to infant in such countries, as the local dental community has neither the financial and physical resources nor the trained dental personnel. We have found an exception to this in the city of Bauru, Sao Paulo, Brazil. This community of 250,000 residents is situated in the sugar cane growing region of Brazil and boasts the leading dental school in South and Central America. In the investigation described, we will collaborate with the Bauru investigators in a longitudinal randomized clinical trial with the following specific aims: 1) to determine whether the salivary levels of the MS can be reduced in mothers of young infants by an intervention program consisting of restorations, topical fluorides, the use of xylitol chewing gum, chlorhexidine varnishes and oral hygiene instructions; 2) to determine whether this intervention reduces or delays the acquisition of MS in the infants and whether this in turn reduces the subsequent caries incidence in children

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Mother
* 20 teeth
* Medically healthy
* First-time mother
* High levels of the mutans streptococci
* No fluoride exposure in the previous 6 months.
* Infant
* Medically healthy
* No cognitive impairment

Ages: 2 Months to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280
Dates: Start 2001-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh-Univesidade de Dao Paulo, Bauru, São Paulo, Brazil